CLINICAL TRIAL: NCT02008487
Title: Novel Wound Powder RGN107 to Reduce Wound Odor, Pain and Exudate at End-of-life
Brief Title: Wound Powder for Pressure Ulcers at End-of-life
Acronym: RGN107
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Teresa Kelechi, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21NR014310 (NIH)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Pressure Ulcer; Wounds
Keywords: wound; palliative care; hospice; pressure ulcers
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries | interventions — RGN107

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Wound powder (Other): In both hospice settings, a registered nurse establishes the wound protocol per principles of wound care and agency guidelines. The cover dressing will be removed and the wound cleansed according to agency protocol (usual care) or as needed. The RGN107 powder, contained in a small squirt bottle, will be squeezed/sprinkled on the wound at each dressing change after cleansing or until a crust is formed. Once formed, the powder will be applied only minimally to reinforce crust integrity. The peri-wound skin will receive care and the cover dressing will be applied. Minimal manipulation of the crusted area will ensue once it has formed. Frequency of dressing changes depends on wound characteristics such as exudate.
  Interventions: Other: Wound powder application

INTERVENTIONS:
Other: Wound powder application — Powder application to wound per protocol.
  Other Names: RGN107; MittiHeal

SUMMARY:
This study will test a special powder for ulcers caused by a variety of conditions such as pressure that sometimes happen when a person is at the end of life. The powder will be applied to these ulcers to see if it helps with pain, odor and drainage (leakage). People who are being cared for by hospice or palliative care organizations will be invited to be in the study. The study will also find out if the powder is easy to use by caregivers as well as improving the comfort and quality of life of the person who has the ulcer.

DETAILED DESCRIPTION:
Aim 1. In a comparative 2-group design, we will evaluate and compare the feasibility of the intervention through assessment in both settings (home-based and inpatient) on:

1. Adherence to RGN107 protocol by licensed care providers and/or family or other caregivers providing wound care; measures include implementation of procedures, frequency of dressing changes.
2. Reach, enrollment, disenrollment, acceptability, satisfaction; measures include difficulties with recruitment and enrollment, side effects such as burning, peri-wound skin irritation.
3. Usability issues such as powder ability to stick to wound and ease of use of applying powder.

Aim 2. Estimate variability of outcome measurements and effect sizes and investigate the presence of a preliminary "signal" of clinical efficacy in two groups of hospice/home health/residential individuals receiving RGN107 in:

1. Physical wound symptoms outcomes, specifically pain, odor and exudate.
2. Quality of life of individuals receiving and caregivers using RGN107.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older
* Patient prognosis > 1 month and < 6 months
* Pressure wounds
* Pain or odor or exudate score > 2 on VAS
* Wound caregiver able to perform required protocol activities

Exclusion Criteria:

* Known allergies to Turmeric, Mint, Sandalwood
* Using negative pressure wound therapy
* Currently using topical creams or ointments applied to wound bed (powder will not adhere to these products)
* Wound with eschar covering (powder will not stick)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
adherence | 4 weeks
  adherence to RGN107 protocol by licensed care providers and/or family or other caregivers providing wound care; measures include implementation of procedures, frequency of dressing changes.
reach | 4 weeks
  reach, enrollment, disenrollment, acceptability, satisfaction; measures include difficulties with recruitment and enrollment, side effects such as burning, peri-wound skin irritation.
usability | 4 weeks
  usability issues such as powder ability to stick to wound and ease of use of applying powder.

SECONDARY OUTCOMES:
symptoms | 4 weeks
  physical wound symptoms outcomes, specifically pain, odor and exudate will be measured with visual analog scales
quality of life | 4 weeks
  quality of life of individuals receiving and caregivers using RGN107.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Roper Hospice, Charleston, South Carolina
  - Hospice of Charleston, North Charleston, South Carolina
  - Odyssey Hospice, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request and findings will be disseminated through publications and presentations.

REFERENCES:
- See also: Information about the study is available to the public at the above site. — http://scresearch.org